CLINICAL TRIAL: NCT03336203
Title: The Impact of Urate-lowering Therapy on Kidney Function in Patients With/Without Gout
Brief Title: The Impact of Urate-lowering Therapy on Kidney Function (IMPULsKF)
Acronym: IMPULsKF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Medical Practice Prof D. Ivanov (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MPIvanov
Record Dates: First submitted 2017-10-07; First posted 2017-11-08 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Gout; CKD Stage 1-4; SUA Level (>8 mg/dL; 480 µmol/L)
Keywords: eGFR, gout, CKD, uric acid, uric acid lowering therapy, hyperuricemia, allopurinol, febuxostat
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — Febuxostat; Tablets; Allopurinol

STUDY DESIGN:
Intervention Model Description: 180 participants in parallel groups. These patients with high SUA level (>8 mg/dL; 480 µmol/L) are going to be divided into 2 arms (90+90) 1) with gout (EULAR's criteria) and 2) without gout but with presence of CKD 1-4)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyperurecemia with gout (Active Comparator): 90 patients with high SUA level (>8 mg/dL; 480 µmol/L) with gout (EULAR's criteria) are going to be treated with allopurinol 300 mg oral tab or febuxostat 80 vg oral tab to achive target SUA levels as 5 mg/dL (300 µmol/L) and ultralow SUA <3 mg/dL (180 µmol/L)
  Interventions: Drug: Febuxostat 80 MG Oral Tablet or Allopurinol 300 MG Oral Tablet
- Hyperurecemia without gout (Active Comparator): 90 patients with high SUA level (>8 mg/dL; 480 µmol/L) withot gout (EULAR's criteria) but with CKD are going to be treated with allopurinol 300 mg oral tab or febuxostat 80 vg oral tab to achive target SUA levels as 5 mg/dL (300 µmol/L) and ultralow SUA <3 mg/dL (180 µmol/L)
  Interventions: Drug: Febuxostat 80 MG Oral Tablet or Allopurinol 300 MG Oral Tablet

INTERVENTIONS:
Drug: Febuxostat 80 MG Oral Tablet or Allopurinol 300 MG Oral Tablet — treatment either with allopurinol or febuxostat

SUMMARY:
This trial aims to investigate the impact of two target levels uric acid-lowering therapy (ULT) caused by hyperuricemia (HU) on kidney function and CKD progression [1] measured by eGFR and albuminuria (A) [2].

The main current tasks include 1) estimation serum uric acid (SUA) level most potential preserving of kidney function 2) the new onset of gouts depending on SUA level, both in gouts' and CKD' objects 3) safety and side effects of target and ultralow SUA levels for evidence-based ULT optimal regime in CKD and non CKD with gout patients. 4) investigation of cardio vascular rick ratio depending on SUA level.

The tasks also include

1. to determine U-curve or directly proportional relationship between SUA and eGFR-EPI in CKD 1-4
2. to evaluate the new onset of goat which depends on SUA level and renal function In this study the optimal ULT for kidney function based on target SUA level in 30 months' treatment with either allopurinol or febuxostat will be determined.

DETAILED DESCRIPTION:
The background and rationale The extended 2016 EULAR updated report states [2] that for patients on ULT, SUA level should be monitored and maintained to <6 mg/dL (360 µmol/L). A lower SUA target (<5 mg/dL; 300 µmol/L) to facilitate faster dissolution of crystals is recommended for patients with severe gout (tophi, chronic arthropathy, frequent attacks) until total crystal dissolution and resolution of gout [5]. SUA level <3 mg/dL (180 µmol/L) is not recommended in the long term. And among EULAR proposals for future research is mentioned the optimal duration for prophylaxis of acute attacks when starting ULT, long-term impact of very low urate levels on the central nervous system, impact of ULT on kidney function.

Since 2013 it has been treating 2 groups of Caucasians adults with gout and with CKD without gout to target SUA level less than <5 mg/dL; 300 µmol/L. The preliminary results had been orally presented at 50th ERA-EDTA Congress (2015) showing that at least 1-year treatment with febuxostat improves GFR and BP control in patients with asymptomatic HU in non-diabetic CKD 2-3. Ultra low SUA target was a benefit with more frequent side effects.

Taking into account the widespread of CKD, gout and availability of ULT it will be reasonable to ascertain the possibilities of allopurinol/febuxostat therapy in these patients. The research planed should be conducted to serve in primary care.

Methods The main concept of this trial is POEM design (Patient Oriented Evidence that Matters) which addresses a widespread clinical problem to primary care physicians as well as nephrologists. This will encounter in their practice uses patient-oriented outcomes which have the potential to change medical practice if the results are valid and applicable.

IMPULsKF is a Clinical Randomized Prospective Controlled Open Multicenter trial that randomly (by chance) assigns 180 participants in parallel groups. These patients with high SUA level (>8 mg/dL; 480 µmol/L) are going to be divided into 2 arms (90+90) 1) with gout (EULAR's criteria) and 2) without gout but with presence of CKD 1-4). There will be 2 target SUA levels in each group as 5 mg/dL (300 µmol/L) and ultralow SUA <3 mg/dL (180 µmol/L) achieved either with allopurinol or febuxostat. The data obtained will be compared with control group (45 with gout without CKD and 45 with CKD).

Ultralow and normal UA level arms are provided concurrent enrolment and follow-up in this groups which will be selected by a random process. The basic study duration is going to be for 36 months including 3 months recruitment period and 3 months post-trial analysis.

The data obtained will be analysed by professional medical statisticians to present eGFR and Albuminuria trends are based on the following: NNT depending target SUA levels, ARR, Likelihood ratio Positive Predictive Value, Odds Ratio and statistical differences between groups comparing Sensitivity and Specificity of both arms treatment.

Primary and secondary outcomes

The primary outcome is comparison benefits of ULT to 2 different targets in

1. Clinical reduction of new onset of acute gout
2. prevention of worsening of kidney function by eGFR measurement
3. estimating CKD prognosis by eGFR and A level The secondary outcomes is comparison benefits of ULT to 2 different targets in

a) cardiovascular risk diminution b) central and peripheral nervous system status c) comparison efficacy, side effects and cost utility between allopurinol and febuxostat d) impact of ACEI/ARB on SUA levels corrected by allopurinol/febuxostat in different CKD stages

Inclusion/exclusion criteria

Inclusion criteria: outpatient adult subjects with hyperurecemia (SUA level above 8 mg/dL (480 µmol/L) either with gout or gout-free CKD 1-4 stages Exclusion criteria: CKD 5, severe forms of associated comorbidities and cardiovascular risk factors, including heart failure III-IV NYHA, stroke, peripheral arterial disease, obesity with BMI above 30 kg/m2, hypertension 3 grade, insulin-dependent DM and any kind of cancer, inpatient intensive unit subjects.

Confounders/covariates.

There are 4 independent centers which will be enrolled to this project.

PI - contract (Shupyk National Medical Academy of Postgraduate Education, location Medical Practice Prof. D.Ivanov)

Subcontract (Liman National Medical University)

Subcontract (SSA "Scientific and Practical Centre of Clinical and Preventive medicine")

Subcontract (Feofaniya Clinical Hospital)

Recruitment/sampling method; sample size calculation (based on WHO recommendations

Participant selection Investigators are inviting the adults with high level of uric acid in blood with or without gout and chronic kidney disease who attend mentioned clinics to participate in the research. No new medicine will be used.

Voluntary Participation

Participation in this research is entirely voluntary. Each patient may change his/her mind later and stop participating even if he/she agreed earlier.

Information on the Trial Drug: allopurinol 300 mg and febuxostat 80-120 mg

These drugs were officially approved in Ukraine for usage in eligibility clinical situation. They had been tested before with people who have elevated uric acid level not successfully controlled by diet. They could be used in patients with gout and CKD. So this research is not the "phase of trial".

Patient could buy this medicine officially in pharmacy for his personal usage according to doctor's prescription. The dosage will be correctly individualized by doctor according to uric acid level and each clinical status.

Procedures and Protocol

First the blood sample will be taken, then according to patient's clinical data and uric acid blood level either allopurinol or febuxostat will be prescribed. In 6 months and every 6 months after uric acid blood level as well as optional biochemistry tests will be performed. During this time patient will have access to his doctor for clinical status monitoring. After 30 months the final exam will be done.

Unfamiliar Procedures Not declared.

Protocol:

1) Involving randomization non-blinded used twice: first for taking either allopurinol or febuxostst, then for achieving target uric acid level.

It is important that neither patient nor doctor know which of the two drugs initially are given. This information will be in investigator's files, but researchers will not look at these files until after the research is finished.

The healthcare workers will be looking after participants very carefully during the study. If doctor are concerned about what the drug is doing, investigator will find out which drug patients are getting and make changes.

If doctor find that the medicine that is being used does not have the desired effect, or not to the extent that he wish it to have, doctor will use "rescue medicine", change the dosage or switch into another one If patient find that the drug are being tested does not stop his/her pain and it is very uncomfortable for him her, so researcher can use the rescue medicine to make patient more comfortable.

The patient will receive the treatment of his condition according to international guidelines.

The researcher will take blood from arm using a syringe and needle. Each time it will be taken about 5 ml of blood. In total, it will be taken about 50 ml in 6 months. At the end of the research, in 3 years, any leftover blood sample will be destroyed.

Description of the Process During the research patient makes 7 visits to the clinic. Following confirmation of contact details and eligibility and after getting informed consent doctor will carry out a health examination, and then draw blood for a laboratory measurement of serum uric acid, creatinine for calculation eGFR-EPI and routine biochemistry tests.

* In the first visit, a small amount of blood, equal to about a teaspoon, will be taken from patient's arm with a syringe. This blood will be tested for the concentration of uric acid. The investigators will also ask patient a few questions about patient's general health and measure how tall he/she is and how much his/her weigh.
* At the next visit, which will be two weeks later, patient will be asked again some questions about his/her health and then he/she will be given either the test drug or the drug that is currently used for decreasing uric acid in patient's blood.
* After 4 week, he/she will come back to the clinic for a blood test. This will clarify drug effect and then his/her visits will every 6 months.

Duration The research takes place over 36 months in total. During that time, it will be necessary for patient to come to the clinic/hospital/ at least 7 days, for 1.5-2 hours each day. The investigators would like to meet with him/her three months after patient's last clinic visit for a final check-up.

In total, patient will be asked to come 8 times (7+1) to the clinic in 30 months. At the end of 30 months, the research will be finished.

Side Effects

As already mentioned, these drugs can have some unwanted effects in low target level. It can make fill pain. It is possible that it may also cause some problems that team are not aware of. However, doctor will follow patient's closely and keep track of any unwanted effects or any problems. Doctor may use some other medicines to decrease the symptoms of the side effects or reactions. Or doctor may stop the use of one or switch from allopurinol to febuxostat or vice versa. If this is necessary doctor should discuss it together with patient and patient will always be consulted before doctor move to the next step.

Risks

By participating in this research it is possible that patient will be at greater risk than he/her would otherwise be. There is, for example, a risk that his/her disease will not get better and that the new medicine doesn't work even as well as the old one. If, however, the medicine is not working and gout signs does not go down in 4 weeks the investigators will individualized the dosage or switch to another one which will make patient more comfortable.

While the possibility of this happening is very low, patient should still be aware of the possibility. Doctor should try to decrease the chances of this event occurring, but if something unexpected happens, doctor will provide patient with medical care he/her needed.

Informed Consent Form Template for Consent for Storage and Future Use is provided.

Statistical methods The data will be entered and analysed using appropriate statistical measures. Categorical data were presented as number and percentage. Continuous data is presented as mean and standard deviation (SD) if normally distributed or median and interquartile range (IQR) if non normal distributed. The Student's t test is used for the comparison of mean and median, respectively. Multiple logistic regression are used for assess the adjusted risk of side effects and cardio-vascular ones. A P value of less than 0.05 is considered to be significant.

Ethical considerations

The study protocol is reviewed by the ethics committee at Shupyk National Medical Academy of Postgraduate Education Kiev, Ukraine. Informed consent to clinical project as well as informed consent for sample storage will be provided.

Reimbursements The investigators and sponsor won't give patient any money or other gifts to take part in this research.

Knowledge translation The data obtained will be presented to ISN as a report and original article and to multidisciplinary medical journal "KIDNEYS" in Ukraine. The final data will be spread to scientific conferences in Ukraine and International meetings. EULAR will be informed about results obtained.

Research team

A multidisciplinary team will ensure the goals of this project are achieved. There are 4 professional centres involves, each of it headed by Prof in Nephrology with rheumatology facilities: Prof Sinjchenko OV, Prof Golovach IYu, Ass Prof Bevzenko TB and Prof Ivanov DD. All centres include departments with well-educated experienced stuff and certificated laboratories and equipment. Unified standardization will be used for all 4 centers. Technical support team will be provided by National Medical Academy of postgraduate education. There are 18 persons in total.

Institutional environment To base the study within the National Medical Academy of Postgraduate Education is perfectly suited to address the needs of the project. It's the largest and most well-experienced organization in clinical projects. However, this study will mainly conduct in 4 principal centres for nephrology and rheumatology care which already have had the experience and preliminary results in this cohort of patients.

Significance

For patients:

If patient participate in this research, he/she will have the following benefits: treatment will be provided according International guidelines to achieve maximum effect for gout and CKD patient probably have had with less side effects; long-time follow-up could give him/her possibility to manage the disease in proper way. There may not be any benefit for patient but his/her participation is likely to help us find the answer to the research question. There may not be any benefit to the society at this stage of the research, but future generations are likely to benefit.

For patients in Ukraine exceptionally. According to our centre every third patient with kidney disease in Ukraine has a level of uric acid more than 420. Choose the right tactics such a patient will have medical and social importance

For specialists:

The investigators are going to answer the following questions:

* do doctor needs to control high uric acid levels in patients with CKD without gout?
* are the new onset of gout depending on SUA level both in gouts' and CKD' objects?
* Which targets are safeties for SUA levels in patients with CKD with gout and without gout?

For ISN and EULAR guidelines:

- the investigators expect to obtain the optimal uric acid lowering therapy practice for preserving renal function based on serum uric acid level in CKD patients with gout/without gout and patients gout without CKD

ELIGIBILITY:
Inclusion Criteria:

* outpatient adults withgout and hyperurecemia (SUA level above 8 mg/dL (480 µmol/L)
* outpatient adults with CKD 1-4 stages and hyperurecemia (SUA level above 8 mg/dL (480 µmol/L)

Exclusion Criteria:

* CKD 5 stage
* heart failure III-IV NYHA
* stroke
* peripheral arterial disease
* obesity with BMI above 30 kg/m2
* hypertension 3 grade
* insulin-dependent DM
* any kind of cancer
* inpatient intensive unit patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2017-10-30 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical reduction of new onset of acute gout attacks | 30 months
  number of attacks
Estimating CKD prognosis by eGFR | 30 months
  eGFR (every 6 months)
Estimating CKD prognosis by Albuminuria | 30 months
  Albuminuria level (every 6 months)

SECONDARY OUTCOMES:
cardiovascular risk diminution | 30 months
  number of all cases of cardiovascular mortality
nervous system status | 30 months
  number of clinical side effects affecting nervous system

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Practice Prof D.Ivanov, Kiev, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided
After finishing trial and results omtained - yes

REFERENCES:
- See also: 2. Richette P, Doherty M, Pascual E, Barskova V, Becce F et al,2016 updated EULAR evidence-based recommendations for the management of gout. Ann Rheum Dis. 2017 Jan;76(1):29-42. doi: 10.1136/annrheumdis-2016-209707. Epub 2016 Jul 25.. — http://dx.doi.org/10.1136/annrheumdis-2016-209707
- See also: 29. Ivanov D. The impact of urate-lowering therapy on kidney function (IMPULsKF). Kidneys, 2017 (6) 2: 91-93.This project aims to investigate the impact of two target levels urate-lowering therapy (ULT) caused by hyperuricemia (HU) on kid — https://doi.org/10.22141/2307-1257.6.2.2017.102786